CLINICAL TRIAL: NCT00664586
Title: A Phase 1 Continuous Intravenous Infusion Study of Terameprocol (EM-1421) in Subjects With Refractory Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding constraints
Sponsor: Erimos Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EM-1421 #104
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Refractory Solid Tumors; Lymphoma
Keywords: Terameprocol (EM-1421); Phase 1; Infusion; Refractory Solid Tumors; Lymphoma; Maximum Tolerated Dose; Tumor Response; Tumor Markers; Pharmacokinetics
MeSH Terms: conditions — Lymphoma | interventions — terameprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Terameprocol (EM-1421) (Experimental): Terameprocol (EM-1421) will be administered as an intravenous infusion over 24 hours, weekly. Dose will commence in the first cohort with 100 mg per hour (2400 mg in a 24 hour period)with escalation in the 5 cohorts of 3 to 6 patients with increments of 25 mg per hour to a maximum of 200 mg/hr (4800 mg/24 hour period) or until MTD is defined. When the MTD has been declared, then 11 additional subjects will be enrolled at the MTD dose level (to total 14 subjects treated in dosage cohort).
  Interventions: Drug: Terameprocol (EM-1421)

INTERVENTIONS:
Drug: Terameprocol (EM-1421) — Weekly (3 of 4 consecutive weeks) 24 hour continuous intravenous infusion
  Other Names: Terameprocol; EM-1421; meso-Tetra-o-Methyl Nordihydroguaiaretic Acid

SUMMARY:
This is a Phase I continuous infusion study designed to explore if constant concentration over time adds to the effectiveness of terameprocol without increasing toxicity. It will also explore weekly dosing as an option.

Tumor response assessments will be performed following every two (2) cycles of therapy. All subjects will undergo a follow-up visit 30 days following their last dose of terameprocol. Circulating tumor cells (CTC) will be quantified pre dosing and on day 15 after first dose of each cycle. Needle biopsy specimens will be taken prior to therapy and one week after first dose, if possible, to assess for tumor markers (cdc-2 and survivin). Tumor markers, for example prostate specific antigen (PSA) will also be measured on day 15 of each cycle (if elevated on study entry). Pharmacokinetic parameters will be derived from analysis of blood samples collected during the first 24 hour infusion.

DETAILED DESCRIPTION:
Subjects meeting all inclusion and exclusion criteria will be enrolled to receive terameprocol as a weekly 24 hour intravenous infusion, three weeks out of four. Serial measurements of safety will be performed prior to dosing. Subjects will be screened within 28 days of Cycle 1. Hematologic, serum chemistry, tumor marker, and pregnancy testing will be performed. Circulating tumor cell assays will be performed. Needle biopsy specimens will be taken prior to therapy and one week after first dose, if possible, to assess for tumor markers (cdc-2 and survivin). Subjects meeting all inclusion and exclusion criteria will be enrolled in groups of 3-6 subjects to receive terameprocol as a weekly 24 hour intravenous infusion. The terameprocol dose levels to be studied include 100mg/hr, increasing by 25 mg/ hr increments in the next cohort assuming no DLT is reached. Serial measurements of safety will be performed at each visit. The MTD will be assessed after the first Cycle of treatment at a dose level. The use of myeloid colony-stimulating factors will not be allowed prophylactically in cycle 1 but may be used if clinically indicated and will be allowed during subsequent cycles to prevent the development of neutropenia in subjects with an established history of this adverse event in earlier cycles. Each subject in a cohort will be treated at the same dose and on the same schedule of weekly infusions. Dose escalation in a subject may be allowed after safe evaluation of a higher dosage, and two cycles being completed with stable disease or better.

Terameprocol (EM-1421) will be administered as an intravenous infusion over 24 hours, weekly. Dose will commence in the first cohort with 100 mg per hour (2400 mg in a 24 hour period)with escalation in the 5 cohorts of 3 to 6 patients with increments of 25 mg per hour to a maximum of 200 mg/hr (4800 mg/24 hour period) or until MTD is defined. When the MTD has been declared, then 11 additional subjects will be enrolled at the MTD dose level (to total 14 subjects treated in dosage cohort).

Cohort A. will receive weekly Terameprocol 100 mg per hour (2400 mg in a 24 hour period)

Cohort B. will receive weekly Terameprocol 125 mg per hour (3000 mg in a 24 hour period)

Cohort C. will receive weekly Terameprocol 150 mg per hour (3600 mg in a 24 hour period)

Cohort D. will receive weekly Terameprocol 175 mg per hour (4200 mg in a 24 hour period)

Cohort E. will receive weekly Terameprocol 200 mg per hour (4800 mg in a 24 hour period)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects greater than or equal to 18 years of age.
2. Subjects who have provided written informed consent to participate in the study.
3. Subjects with documented evidence of cancer with clinically measurable or evaluable disease. Cancer can be recurrent after primary treatment with surgery, radiation therapy and/or chemotherapy and may include those subjects for whom no standard or curative therapy exists.
4. Measurable tumor by imaging (CT per RECIST criteria). unless an established tumor marker exists which can be used for assessment of response in the absence of measurable disease (i.e., PSA in prostate cancer or CA 125 in ovarian cancer).
5. No recent myocardial infarction (within 3 months) or serious intercurrent cardiovascular disease (any event that requires evaluation by a cardiologist, with a definitive cardiac disease diagnosed) Subjects with a history of severe cardiac disease should have had a recent consultation with a cardiologist documenting that there are no new findings.
6. No overt cardiac metastasis.
7. Negative pregnancy test if in women of childbearing potential within one week of starting therapy.
8. ECOG Performance Status of 0, 1, or 2.
9. Absolute neutrophil greater than or equal to 1500 cells/uL, hemoglobin greater than or equal to 9 gm/dl, platelets greater than or equal to 100,000/uL, ALT/AST less than or equal to 3 x ULN (upper limit of the normal range) unless involved with tumor then less than 5 x ULN, bilirubin less than or equal to 1.5 x ULN, creatinine less than or equal to 1.5 x ULN, normal creatinine clearance greater than 60 mL/min and a normal serum bicarbonate. Normal is defined by local laboratory specifications.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be considered eligible for participation in the study:

1. Women who are pregnant or breast-feeding (women of child-bearing potential must have a negative serum pregnancy test within one week of entering the study).
2. Women of child-bearing potential who are unwilling to use two medically acceptable forms of contraception during the course of the study (surgical sterilization, approved hormonal contraceptives, or barrier method with spermicide).
3. Subjects unable to comply with the study requirements.
4. Subjects with a known sensitivity to any of the study medication components.
5. Subjects exhibiting any of the following: a marked baseline prolongation of QT/QTc interval (repeated demonstration of a calculated QTc interval >450), a history of additional risk factors for TdP (e.g. heart failure, hypokalemia, family history of long QT Syndrome), and subjects unable or unwilling to refrain from using medications that are known to prolong the QT/QTc ratio during the course of the study. Subjects having recently taken such medications must have five half-lives off medication before participation.
6. Subjects with an existing port not compatible with the terameprocol formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine Maximum Tolerated Dose (MTD)and dose limiting toxicities (DLTs) of Terameprocol (EM-1421) administered as a weekly continuous infusion over 24 hours. | The MTD will be assessed after the first Cycle of study drug treatment

SECONDARY OUTCOMES:
To further assess the anti-tumor activity of intravenously administered Terameprocol using objective response and duration of response. | Subjects will be evaluated for response after every 2 cycles (8 weeks) while on study drug.
To assess the pharmacokinetic parameters Terameprocol administered as 24 hour intravenous infusions. | Pharmacokinetics samples will be taken on Day 1 only: pre-dose and at 1, and 4 hours, 24 hours, 25 hours and 26 hours after first study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Frazer, MB, ChB, Study Director — Erimos Pharmaceuticals
Locations (1):
- The Sarah Cannon Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related information — http://www.erimos.com